CLINICAL TRIAL: NCT06423911
Title: This is a Global, Multi-center, Open-label Randomized and Registrational Phase 3 Study of Olverembatinib (HQP1351) in Patients With Chronic Phase Chronic Myeloid Leukemia
Brief Title: Study of Olverembatinib (HQP1351) in Patients With CP-CML
Acronym: POLARIS-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351CG301
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Myeloid Leukemia; CML; CML, Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — olverembatinib; bosutinib

STUDY DESIGN:
Intervention Model Description: Part A 2:1 ratio Part B: control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A, RCT, olverembatinib arm and bosutinib arm (Other): Randomized controlled part that is designed to compare the efficacy and safety of olverembatinib (investigational arm) versus bosutinib (control arm) in patients with CML-CP, previously treated with at least two TKIs
  Interventions: Drug: olverembatinib; Drug: Bosutinib
- Part B, SAT, olverembatinib arm (Other): To evaluate the efficacy and safety of olverembatinib in the CML-CP patients with T315I mutation previously
  Interventions: Drug: olverembatinib

INTERVENTIONS:
Drug: olverembatinib — olverembatinib QOD
Drug: Bosutinib — Bosutnib QD
  Arms: Part A, RCT, olverembatinib arm and bosutinib arm

SUMMARY:
A Global Multicenter, Open Label, Randomized, Phase 3 Registrational Study of Olverembatinib (HQP1351) in Patients with Chronic Phase Chronic Myeloid Leukemia (POLARIS-2)

DETAILED DESCRIPTION:
The hypothesis suggests that in Part A, olverembatinib leads to a higher MMR rate compared to bosutinib in CP-CML patients without the T315I mutation; and in Part B, olverembatinib can provide therapeutic benefits to CP-CML patients with the T315I mutation.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all of the following criteria.

1. Age ≥ 18 years old.
2. Diagnosis of CML-CP
3. Part A: Previously treated with at least two approved TKIs Part B: T315I mutation at screening.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
5. Written informed consent obtained prior to any screening procedures.
6. Patients with adequate organ functions

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria.

1. For Part A only: T315I mutation at any time prior to starting study treatment.
2. Active infection that requires systemic drug therapy
3. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter absorption of study drugs
4. Previous treatment with or known / suspected hypersensitivity to olverembatinib or any of its excipients.
5. Previous treatment with or known / suspected hypersensitivity to bosutinib or any of its excipients.
6. Pregnant or nursing (lactating) women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MMR rate Part A | 24 weeks
  To compare the major molecular response (MMR) rate at 24 weeks of olverembatinib versus bosutinib
MMR rate Part B | 24 weeks
  To evaluate the MMR rate by 24 weeks of olverembatinib in CML-CP patients with T315I mutation

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States